CLINICAL TRIAL: NCT00265239
Title: Effects of Edaravone in Patients With Acute Myocardial Infarction
Brief Title: Pilot Study of Edaravone to Treat Acute Myocardial Infarction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kumamoto University (Other)
Collaborators: Japan Heart Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 310
Record Dates: First submitted 2005-12-13; First posted 2005-12-14 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2007-11

CONDITIONS: Myocardial Infarction; Reperfusion Injury
Keywords: Edaravone; Randomized Control Trial; ST-Elevation Myocardial Infarction; Coronary Angioplasty
MeSH Terms: conditions — Myocardial Infarction; Reperfusion Injury; ST Elevation Myocardial Infarction | interventions — Edaravone

ARMS (2):
- 1 (Active Comparator): Edaravone Group
  Interventions: Drug: edaravone
- 2 (No Intervention): Placebo Group

INTERVENTIONS:
Drug: edaravone — intravenous administration of 30mg Edaravone just before reperfusion therapy
  Arms: 1

SUMMARY:
Early reperfusion therapy has improved the clinical outcomes of patients with acute myocardial infarction (AMI), but these benefits are limited in some patients by reperfusion injuries. There is now increasing evidence that reactive oxygen species cause reperfusion injury. This study was designed to examine the effects of edaravone, a novel free radical scavenger, in patients with AMI.

DETAILED DESCRIPTION:
Initial AMI patients were randomly assigned to receive 30 mg of edaravone or a placebo intravenously just before reperfusion. We compared infarct size, using serial determination of serum biomarkers and Q wave formations, and the incidence of reperfusion arrhythmia between the groups. Cardiovascular event-free curves were estimated by Kaplan-Meier method. In addition, we determined serum thioredoxin levels, an oxidative stress marker, to assess the antioxidant effect of edaravone.

ELIGIBILITY:
Inclusion Criteria:

* Initial AMI patients admitted to the investigators' institution within 6 hours of symptom onset and treated primary percutaneous coronary intervention.

Exclusion Criteria:

* Renal insufficiency defined as serum creatinine > 1.2 mg/dl and altered hepatic function defined as serum asparate aminotransferase > 50 IU/L, alanine aminotransferase > 50 IU/L and total bilirubin > 1.2 mg/dl.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2001-04; Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hisao Ogawa, MD, PhD, Study Chair — Department of Cardiovascular Medicine, Graduate School of Medical Sciences, Kumamoto University
Locations (1):
- Department of Cardiovascular Medicine, Graduate School of Medical Sciences, Kumamoto University, Kumamoto, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- Edaravone Group: Edaravone Group
  edaravone: intravenous administration of 30mg Edaravone just before reperfusion therapy
- Placebo Group: Placebo Group
Period: Overall Study
Arm/Group | Edaravone Group | Placebo Group
Started | 52 | 52
Completed | 50 | 51
Not Completed | 2 | 1
Not completed — Adverse Event | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Edaravone Group | Placebo Group | Total
Number analyzed (Participants) | 50 | 51 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (2) | 63 (2) | 63 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 16 | 26
  Male | 40 | 35 | 75
Region of Enrollment [Number; unit: participants]
  Japan | 50 | 51 | 101

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Death
Description: number of cardiac death
Time Frame: 415±32 days
Measure: Number; unit: events
Arm/Group | Edaravone Group | Placebo Group
Number analyzed (Participants) | 50 | 51
events | 0 | 0

2. Primary Outcome: Nonfatal Myocardial Reinfarction
Description: number of nonfatal myocardial reinfarction
Time Frame: 415days
Measure: Number; unit: events
Arm/Group | Edaravone Group | Placebo Group
Number analyzed (Participants) | 50 | 51
events | 0 | 2

3. Primary Outcome: Refractory Angina Pectoris
Description: number of refractory angina pectoris
Time Frame: 415days
Measure: Number; unit: events
Arm/Group | Edaravone Group | Placebo Group
Number analyzed (Participants) | 50 | 51
events | 1 | 5

4. Primary Outcome: Nonfatal Ischemic Stroke
Description: number of nonfatal ischemic stroke
Time Frame: 415days
Measure: Number; unit: events
Arm/Group | Edaravone Group | Placebo Group
Number analyzed (Participants) | 50 | 51
events | 0 | 1

ADVERSE EVENTS:
Description: adverse events were only collected during the therapy period, up to 2 weeks
Arm/Group | Edaravone Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/51
Other Adverse Events (participants affected / at risk) | 0/50 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes